CLINICAL TRIAL: NCT06889077
Title: The Effect of QR Code-Supported Perioperative Education Material Used in Clinical Practice on Nursing Students Knowledge Levels and Attitudes Towards Evidence-Based Practices: a Randomised Controlled Trial
Brief Title: The Effect of QR Code-Supported Perioperative Education Material Used in Clinical Practice
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Emine Arici Parlak, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15151515
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Clinical Practice; Nursing Education; Nursing Students; Evidence Based Nursing
Keywords: Clinical Practice; Nursing Students; Nursing Education; Evidence Based Nursing; Knowledge Level; Quick Response Code

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QR Code Group (Experimental): Students will receive support in their clinical practice through QR Code-supported perioperative education materials.
  Students knowledge level and attitudes towards evidence-based nursing will be evaluated after clinical practice.
  Interventions: Other: QR Code Group
- Control Group (No Intervention): Students knowledge level and attitudes towards evidence-based nursing will be evaluated after clinical practice.

INTERVENTIONS:
Other: QR Code Group — Students will receive support in their clinical practice through QR Code-supported perioperative education materials.
  Arms: QR Code Group

SUMMARY:
This study is planned as a randomized controlled trial to examine the effects of the use of QR (Quick Response) Code-supported materials prepared for perioperative care by nursing students during clinical practice on the knowledge levels of nursing students and their attitudes towards evidence-based nursing.

DETAILED DESCRIPTION:
Evidence-based nursing is an approach that started with the works of Florence Nightingale and aims to base nursing practices on scientific foundations over time. Nurses must have a variety of roles, including the roles of caregiver, educator, leader, and patient advocate, as well as a commitment to evidence-based practice. Therefore, instead of traditional learning methods, students should learn evidence-based practices and take on roles during their clinical practice to provide safe and high-quality care in order to have a professional identity professionally. The World Health Organization (2016) report on "Nurse Educator Core Competencies" recommends that nurse educators facilitate active learning in the education process, select and use appropriate technologies and materials, and encourage individualized experiential learning. For this reason, in addition to constantly innovative health practices, new developments in the field of educational technologies should be followed closely. QR (Quick Response) Code technology is a tool used to share web-based information. The use of QR Codes in education is an innovative approach. It makes the education process of nursing students interactive with today's technology and increases student participation and access to education.

Upon reviewing the literature, no studies were found that evaluated the effect of QR Code-supported education, which is an innovative education method in nursing students during clinical practice, on the students' knowledge level and evidence-based attitude. Therefore, this study is planned to be conducted on nursing students. The results of this study are expected to contribute to that students will participate interactively in the evidence-based learning and practicing process during clinical education, and the educational methods used will gain a critical and innovative approach for both students and educators.

The study will conduct as a prospective randomized controlled trial. After obtaining verbal and written consent from the students before and after the clinical practice, the study will conduct with various data collection forms.

These forms are; Student Identification Form, Knowledge Level Measurement Test for Evidence-Based Practices Including Perioperative Care, Evidence-Based Nursing Attitude Questionnaire, Form for Opinions on the Use of QR Codes will be used.

The QR (Quick-Response) group in group- I (n=30), and group II (n=30) will be the control group. The study has 2 stages. In the first stage, the descriptive characteristics of the participants and their knowledge level regarding evidence-based practices including perioperative care will be measured for both groups.

During the second stage of their clinical practice, participants in the intervention group will receive support through QR code-enabled perioperative educational materials. These QR code-supported resources will be available to the participants throughout their entire clinical education process. Participants in the control group will continue their clinical practice using the learning methods available in the educational curriculum. Following clinical practice with participants in both intervention and control groups, researchers will assess participants' knowledge levels using a measurement test focusing on evidence-based practices including perioperative care. Additionally, participant's attitudes toward evidence-based nursing will be assessed using an attitude scale on this topic. In addition, researchers will collect participants' opinions on using QR Codes in the intervention group through a designated feedback form.

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year student at Gülhane Nursing Faculty of Health Sciences University
* Agreeing to participate in the study

Exclusion Criteria:

* Not completing any stage of the study
* Wanting to withdraw from the study
* Having previously taken the surgical disease nursing course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Having taken a course in surgical diseases nursing
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Change from knowledge level in clinical practice | After Using QR Codes in Clinical Practice. An average of 5 months.
  Educational materials supported by QR codes will enhance students' knowledge of perioperative care in clinical practice. This status will be assessed through a Post-Test measuring knowledge of evidence-based practices in perioperative care. The Post-Test, developed by the researchers, consists of 20 questions, each with four answer options. Each correct answer is worth 5 points, resulting in a possible score range from 0 to 100. A higher score indicates a greater level of knowledge.

SECONDARY OUTCOMES:
Changes in attitude toward evidence-based nursing after clinical practice | After Using QR Codes in Clinical Practice. An average of 5 months.
  Participants' use of QR Codes during the clinical practice process will affect their attitudes towards evidence-based nursing. This status will be evaluated with the Attitude Scale towards Evidence-Based Nursing. The Attitude Scale towards Evidence-Based Nursing consists of 15 items and 3 sub-dimensions. The total score is 15-75. A high score on the scale indicates a positive attitude towards evidence-based nursing. (Ruzafa-Martínez et al. 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Emine Arici Parlak, PhD, Principal Investigator — University of Health Sciences Turkiye Gulhane Faculty of Nursing
Locations (1):
- University of Health Sciences Turkiye Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)